CLINICAL TRIAL: NCT02238444
Title: Efficacy and Safety of Warfarin Anticoagulation for Prevention of Portal Vein Thrombosis in Liver Cirrhotic Patients With Hypersplenism After Laparoscopic Splenectomy
Brief Title: Warfarin Prevents Portal Vein Thrombosis in Liver Cirrhotic Patients With Hypersplenism After Laparoscopic Splenectomy
Acronym: ESWA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Master, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YZUC-001
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Cirrhosis; Hypertension; Venous Thrombosis; Status; Splenectomy
Keywords: Warfarin; Portal Vein; Anticoagulants; Cirrhosis; Hypertension; Venous Thrombosis; Splenectomy
MeSH Terms: conditions — Fibrosis; Hypertension; Venous Thrombosis | interventions — Warfarin; Dipyridamole; Aspirin; aspirin, magnesium oxide combination; Heparin, Low-Molecular-Weight; Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warfarin with dipyridamole (Experimental): From postoperative day 3, patients will receive dipyridamole 25mg tid for three months along with subcutaneous Low Molecular Weight Heparin Calcium injection for first five days and Warfarin 2.5mg qd with titration of dose to maintain a target INR of 2-3. Intially the INR will be monitored twice weekly with gradual escalation of dose to achieve target INR. After achieving the target INR, this is to be repeated every 4 weeks. The Doppler Ultra Sonography screening will be done every 3 months to assess the occurrence of portal vein thrombus, but the medications will be continue for one year irrespective of the occurrence of portal vein thrombus.
  Interventions: Drug: Warfarin; Drug: Dipyridamole; Drug: Low Molecular Weight Heparin
- Aspirin with dipyridamole (Active Comparator): From postoperative day 3, patients will receive oral dipyridamole 25mg tid for three months along with subcutaneous injection of Low Molecular Weight Heparin (4100 IU) for first five days and Aspirin Enterie Ccoated Tablets 100mg qd for one year.
  Interventions: Drug: Dipyridamole; Drug: Aspirin; Drug: Low Molecular Weight Heparin

INTERVENTIONS:
Drug: Warfarin — From postoperative day 3, patients will receive oral Warfarin 2.5mg qd with titration of dose to maintain a target INR of 2-3 for 1 year.
  Other Names: Warfarin Sodium; Athrombine; COUMADIN; PANAWARFIN
  Arms: Warfarin with dipyridamole
Drug: Dipyridamole — From postoperative day 3, patients will receive oral dipyridamole 25mg tid for three months.
  Other Names: Gardoxin; Coribon; Curantyl; Dilaplus
Drug: Aspirin — From postoperative day 3, patients will receive oral Aspirin Enterie Ccoated Tablets 100mg qd for 1 year.
  Other Names: Acenterine; Acetard; Acetophen
  Arms: Aspirin with dipyridamole
Drug: Low Molecular Weight Heparin — From postoperative day 3, Patients will receive subcutaneous injection of Low Molecular Weight Heparin (4100 IU) once daily for first five days.
  Other Names: Fraxiparine

SUMMARY:
The purpose of this study is to determine whether Warfarin Anticoagulation are effective and safe in Prevention of Portal Vein Thrombosis in Liver Cirrhotic Patients with Hypersplenism after Laparoscopic Splenectomy.

DETAILED DESCRIPTION:
After successful screening the cases of cirrhosis of liver irrespective of the etiology who have non tumor portal vein thrombosis will be enrolled. The baseline Doppler parameter will be recorded and the patient will be randomized into either interventional (warfarin) or control (aspirin) group. From postoperative day 3, patients in interventional (warfarin) group will receive oral Warfarin 2.5mg qd with titration of dose to maintain a target INR of 2-3 for 1 year, patients in control (aspirin) group will receive oral Aspirin Enterie Ccoated Tablets 100mg qd for 1 year, and both groups will be along with five days of subcutaneous injection of Low Molecular Weight Heparin and three months of oral Dipyridamole. Every 3 months the Doppler screening for the occurrence of portal vein thrombus (PVT) or spleno-mesenteric thrombosis will be done for all patients. Both groups will receive the therapy for one year irrespective of the Doppler findings in relation to portal vein thrombus occurrence. Then one year monitoring will be done in the both groups as per the primary or secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis of any etiology
* Splenomegaly with secondary hypersplenism, Platelet count < 50*10^9/L
* No evidence of PVT or spleno-mesenteric thrombosis by ultrasound evaluation and angio-CT
* Informed consent to participate in the study

Exclusion Criteria:

* Hepatocellular carcinoma or any other malignancy
* Hypercoagulable state other than the liver disease related
* DRUGS- oral contraceptives, anticoagulation or anti-platelet drugs
* Base line INR >2
* Child-Pugh grade C
* Recent peptic ulcer disease
* History of Hemorrhagic stroke
* Pregnancy
* Uncontrolled Hypertension
* Age>75 yrs
* F2 varices with red whale marks or F3 varices
* Bleeding portal hypertension
* Human immunodeficiency virus (HIV) infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09-01; Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportions of patients who will suffer from PVT or spleno-mesenteric thrombosis between oral anticoagulant Warfarin with dipyridamole group and oral Aspirin with dipyridamole group during the study period of 3 year from randomization | 3 years

SECONDARY OUTCOMES:
Proportions of patients who will show improvement in Child Pugh (>2 points)in both groups | 3 years
Proportions of patients who will show improvement in Model for End Stage Liver Disease (MELD)(>4 points)in both groups | 3 years
Proportions of patients who will show decrease in hepatic decompensation defined as development of ascites, PSE, portal hypertensive bleeding, jaundice, spontaneous bacterial peritonitis, or systemic infection | 3 years
Proportions of patients who will suffer from hepatocellular carcinoma | 3 years
Overall survival in both groups | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dou-Sheng Bai, MD, Study Chair — Clinical Medical College of Yangzhou University; Guo-Qing Jiang, MS, Study Director — Clinical Medical College of Yangzhou University; Ping Chen, MD, Principal Investigator — Clinical Medical College of Yangzhou University; Sheng-Jie Jin, Principal Investigator — Clinical Medical College of Yangzhou University
Locations (1):
- Clinical Medical College of Yangzhou University, Yangzhou, Jiangsu, China